CLINICAL TRIAL: NCT03193671
Title: Evaluation and Implementation of New Biomarkers and Algorithms for Diagnosis of Ovarian Cysts/Tumors in the Pelvis
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Karin Sundfeldt, Professor, Göteborg University
Other Study IDs: Ksundfeldt
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Neoplasms; Diagnoses Disease; Biomarkers; Algorithms
Keywords: HE4; CA125; RMI; ROMA
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Benign: Benign tumors, pre-and postmenopausal
  Interventions: Diagnostic Test: Diagnosis
- Malignant: Malignant tumors, pre-and postmenopausal
  Interventions: Diagnostic Test: Diagnosis
- Borderline: Borderline tumors, pre-and postmenopausal
  Interventions: Diagnostic Test: Diagnosis
- Malignant+borderline: Malignant+borderline tumors, pre-and postmenopausal
  Interventions: Diagnostic Test: Diagnosis

INTERVENTIONS:
Diagnostic Test: Diagnosis — Improving diagnosis

SUMMARY:
This study evaluates the biomarkers CA125 and HE4 and the algorithms RMI and ROMA on a normal population in the western region of Sweden. The aim is to improve diagnosis of ovarian cancer.

If the investigators observe a clear improvement in the early diagnosis of EOC, the investigators aim to implement the best strategy for all patients with suspected pelvic tumor mass in the western region of Sweden.

DETAILED DESCRIPTION:
The investigators are currently using CA125 and RMI in diagnosing patients with a pelvic cyst/tumor and referring them to tertiary centers for surgery in the western region of Sweden. The diagnostic accuracy is unsatisfying why the investigators are evaluating HE4 and ROMA as a complement, in combination or separately to improve diagnostic accuracy.

The trial is based on a normal population cohort of patients included at all the hospitals in the region. The patients were included before surgery and the biomarkers analysed on serum samples withdrawn preoperatively.

If the investigators observe a clear improvement in the early diagnosis of EOC, the investigators aim to implement the best strategy for all patients with suspected pelvic tumor mass in the western region of Sweden.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, understand spoken and written Swedish information, admitted for surgery for a cyst/tumos in the pelvis

Exclusion Criteria:

* Rejected participation, cytotoxic chemotherapy prior to surgery, rejected surgery, serum sample failure, already included at another hospital

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on gender identity
Study Population: Patients diagnosed with a cyst/tumor in the pelvis already enrolled for surgery. Included at 6 different Hospitals.
Sampling Method: Probability Sample
Enrollment: 684 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Can the investigators improve diagnostic accuracy in women diagnosed with a cyst/tumor in the pelvis | 12 months
  Finding the true cases and avoiding unnecessary surgery, a descriptive analysis of a normalpopulation

SECONDARY OUTCOMES:
Improve triage of patients to tertiary centers for surgery | 12 months
  Referring the correct cases from a normal population.

CONTACTS AND LOCATIONS:
Locations (1):
- Gothenburg University, Sahlgrenska University Hospital, Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
All IPD are coded with a unique number only available to the main researchers

REFERENCES:
- [Derived] Lycke M, Ulfenborg B, Malchau Lauesgaard J, Kristjansdottir B, Sundfeldt K. Consideration should be given to smoking, endometriosis, renal function (eGFR) and age when interpreting CA125 and HE4 in ovarian tumor diagnostics. Clin Chem Lab Med. 2021 Aug 13;59(12):1954-1962. doi: 10.1515/cclm-2021-0510. Print 2021 Nov 25. PMID 34388324